CLINICAL TRIAL: NCT04077658
Title: A Pilot Single-center Randomized Controlled Study of the Effects of Smartphone Based Heart Rate Variability Biofeedback in People With Migraine
Brief Title: Heartmath Migraine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-00479
Record Dates: First submitted 2019-08-19; First posted 2019-09-04 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Migraine
Keywords: HeartMath app; Inner Balance Sensor
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with intervention arm and waitlist control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeartMath (Experimental)
  Interventions: Behavioral: HeartMath
- Waitlist Control (Active Comparator)
  Interventions: Behavioral: HeartMath; Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: HeartMath — HeartMath is a program where individuals learn heart rate variability biofeedback. Essentially, they learn breathing exercises that reduce their heart rate. The HeartMath program will be administered via an application on the smartphone and ear monitor.
Behavioral: Waitlist Control — Standard of Care Migraine Treatment
  Arms: Waitlist Control

SUMMARY:
This is a two arm study comparing smartphone based heart rate variability biofeedback using the HeartMath app and InnerBalance sensor to waitlist control on migraine quality of life.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether there is any superiority between an 8-week program of app based HRV biofeedback (HeartMath) compared to wait list control in migraine quality of life. Investigators will also look:

* To determine whether there is any superiority between an 8-week program of app based HRV biofeedback (HeartMath) and wait list control in depression in people with migraine.
* To determine whether there is any superiority between an 8-week program of app based HRV biofeedback (HeartMath) and wait list control in anxiety in people with migraine.
* To determine whether there is any superiority between an 8-week program of app based HRV biofeedback (HeartMath) and wait list control in insomnia in people with migraine.

ELIGIBILITY:
Inclusion Criteria:

* International Classification of Headache Disorders (ICHD) 3 criteria for migraine
* 4-20 headache days/month
* Has not done behavioral therapy for migraine in the past year
* Has a smartphone and willing to try HRV biofeedback using an app and ear monitor
* English speaking
* HS graduate or higher level of education
* Patients must not make preventive medication changes for the course of the study. If patients just changed their preventive medication, they must wait a month before enrolling.

Exclusion Criteria:

* Doing any form of behavioral therapy for pain in the past year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
To determine whether there is any superiority between an 8-week program of app based HRV biofeedback (HeartMath) compared to wait list control in migraine quality of life | 8 Weeks
  Measured by comparing the slope of reduction in MSQv2 scores

SECONDARY OUTCOMES:
Change in depression | 8 Weeks
  Measured using slope in reduction of Generalized Anxiety Disorder 7-item (GAD-7) scale. Average scores of 5-9: Mild; 10*-14:Moderate; >15:Severe
Change in anxiety | 8 Weeks
  Measured using slope of reduction in eight-item Patient Health Questionnaire depression scale (PHQ-8), The PHQ-8 uses a 4-point Likert scale to assess depressive symptoms. The score range is 0 to 27. Scores 5-9 indicate "mild" symptoms, 10-14 "moderate", and ≥20 "severe" depressive symptoms.
Change insomnia | 8 Weeks
  Measured using slope of reduction in Insomnia Severity Index (ISI). The ISI is a 7-item questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance, early morning awakening problems; sleep dissatisfaction; interference of sleep problem with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale (0-4) is used to rate each item, yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, MPH, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Mia.Minen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.